CLINICAL TRIAL: NCT02288364
Title: Does Sodium Bicarbonate Reduce the Pain of Lidocaine for Local Anesthesia in Percutaneous Breast Biopsies?
Brief Title: Reducing Pain of Lidocaine Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Pro00056728
Record Dates: First submitted 2014-10-13; First posted 2014-11-11 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-02

CONDITIONS: Pain of Anesthesia at Breast Biopsy
MeSH Terms: interventions — Lidocaine; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1% Lidocaine (Active Comparator): 1% Lidocaine alone.
  Interventions: Drug: 1% Lidocaine
- 1% Lidocaine plus sodium bicarbonate (Active Comparator): 1% Lidocaine plus 8.4% sodium bicarbonate
  Interventions: Drug: 1% Lidocaine plus sodium bicarbonate

INTERVENTIONS:
Drug: 1% Lidocaine
  Arms: 1% Lidocaine
Drug: 1% Lidocaine plus sodium bicarbonate
  Arms: 1% Lidocaine plus sodium bicarbonate

SUMMARY:
The purpose of this study is to determine the benefit, if any, of buffering lidocaine (adding sodium bicarbonate) when used for local anesthesia prior to percutaneous breast needle core biopsies. The medicine doctors use to reduce the pain of breast biopsies, lidocaine, can cause pain for approximately 15 seconds until the numbing effect begins. It is possible that this pain is caused because lidocaine is acidic. Some physicians believe that reducing the acidity of lidocaine by mixing it with sodium bicarbonate will reduce the initial pain of injecting the lidocaine. Both approaches - injecting 1% lidocaine alone and injecting 1% lidocaine mixed with sodium bicarbonate - are used as routine standard of care by radiologists today. The purpose of this study is to determine if either approach is more comfortable for patients having breast procedures.

ELIGIBILITY:
Inclusion Criteria:

* 21 Years of age
* Any patient scheduled for a breast biopsy at Duke Breast Interventional Imaging

Exclusion Criteria:

* Less than 21 Years of age
* Allergic to Lidocaine or Sodium Bicarbonate
* Not mentally capable of consenting

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay A Baker, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 88 participants signed consent. 86 participants were randomized.
Period: Overall Study
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate
Started | 42 | 44
Completed | 42 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.26 (13.70) | 53.80 (13.22) | 53.53 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 44 | 86
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 28 | 31 | 59
  Black | 11 | 13 | 24
  Asian | 2 | 0 | 2
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 42 | 44 | 86

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: Measure of pain on a scale of 0-10. Zero would indicate no pain while a score of 10 would be the worse pain possible.
Time Frame: immediately prior to anesthetizing, within approximately 1 minute of starting
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate
Number analyzed (Participants) | 42 | 44
units on a scale | 1.19 (1.92) | 0.56 (1.30)

2. Secondary Outcome: Pain
Description: Measure of pain on a scale of 0-10. Zero would indicate no pain while a score of 10 would be the worse pain possible.
Time Frame: immediately on completion of anesthetizing the skin, within approximately 1 minute of starting
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate
Number analyzed (Participants) | 42 | 44
units on a scale | 2.07 (2.05) | 1.61 (1.99)
Statistical Analysis 1: Comparison: 1% Lidocaine vs 1% Lidocaine Plus Sodium Bicarbonate; Test type: Superiority or Other; p = 0.30, Chi-squared

3. Secondary Outcome: Pain
Description: Measure of pain on a scale of 0-10. Zero would indicate no pain while a score of 10 would be the worse pain possible.
Time Frame: immediately on completion of anesthetizing the parenchyma (deeper breast tissue), within approximately 4 minutes of starting
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate
Number analyzed (Participants) | 42 | 44
units on a scale | 2.98 (2.67) | 2.02 (2.37)
Statistical Analysis 1: Comparison: 1% Lidocaine vs 1% Lidocaine Plus Sodium Bicarbonate; Test type: Superiority or Other; p = 0.08, Chi-squared

4. Secondary Outcome: Pain
Description: Measure of pain on a scale of 0-10. Zero would indicate no pain while a score of 10 would be the worse pain possible.
Time Frame: immediately on completion of the biopsy, within approximately 20 minutes of starting
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate
Number analyzed (Participants) | 42 | 44
units on a scale | 1.45 (2.65) | 0.91 (2.06)
Statistical Analysis 1: Comparison: 1% Lidocaine vs 1% Lidocaine Plus Sodium Bicarbonate; Test type: Superiority or Other; p = 0.29, Chi-squared

5. Secondary Outcome: Pain
Description: Measure of pain on a scale of 0-10. Zero would indicate no pain while a score of 10 would be the worse pain possible.
Time Frame: 30 seconds after initiating superficial injection in the subcutaneous tissue, within approximately 1 minute of starting
Population: Data not collected at this time point.
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Pain
Description: Measure of pain on a scale of 0-10. Zero would indicate no pain while a score of 10 would be the worse pain possible.
Time Frame: immediately prior to injection of "deep" anesthesia in the breast parenchyma, within approximately 4 minutes of starting
Population: Data not collected at this time point.
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pain
Description: Measure of pain on a scale of 0-10. Zero would indicate no pain while a score of 10 would be the worse pain possible.
Time Frame: 30 seconds after initiating deep injection of the parenchyma (deeper breast tissue), within approximately 4 minutes of starting
Population: Data not collected at this time point.
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Pain
Description: Measure of pain on a scale of 0-10. Zero would indicate no pain while a score of 10 would be the worse pain possible.
Time Frame: immediately prior to obtaining the first core biopsy specimen, within approximately 15 minutes of starting
Population: Data not collected at this time point.
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Pain
Description: Measure of pain on a scale of 0-10. Zero would indicate no pain while a score of 10 would be the worse pain possible.
Time Frame: immediately after obtaining the first core biopsy specimen, within approximately 15 minutes of starting
Population: Data not collected at this time point.
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Pain
Description: Measure of pain on a scale of 0-10. Zero would indicate no pain while a score of 10 would be the worse pain possible.
Time Frame: immediately on completion of the final core biopsy specimen, within approximately 20 minutes of starting
Population: Data not collected at this time point.
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | 1% Lidocaine | 1% Lidocaine Plus Sodium Bicarbonate
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/44
Other Adverse Events (participants affected / at risk) | 0/42 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes